CLINICAL TRIAL: NCT05907018
Title: Comparing Phenotypic and Autonomic Physiologic Determinants of Neurocardiogenic Syncope
Brief Title: Autonomic Monitoring in Neurocardiogenic Syncope
Acronym: ANSS
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0841
Record Dates: First submitted 2023-05-23; First posted 2023-06-18 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Syncope; Chest Pain; Dyspnea
MeSH Terms: conditions — Syncope; Chest Pain; Dyspnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective observational pilot study of suitability of autonomic monitoring via the VU-AMS device for prediction of neurocardiogenic syncope (NCS) in children referred to cardiopulmonary exercise testing (CPET) for a diagnosis of syncope. The study population is children referred for CPET to evaluate for neurocardiogenic syncope. The purpose is to describe autonomic function during rest and exercise and determine the positive predictive value of autonomic function measurements against the gold standard for diagnosis of neurocardiogenic syncope, the CPET. Children presenting for CPET with chest pain or who are status post orthotopic heart transplantation will serve as positive and negative controls respectively.

ELIGIBILITY:
Inclusion Criteria:

* Parent/Legal guardian able to provide informed consent
* Verbal participant assent
* Undergoing clinically indicated CPET.
* Diagnosis of either syncope, chest pain/dyspnea or status post OHT
* Participant willing and able to participate in study procedures
* Age 7-24 years

Exclusion Criteria:

* Participant unwilling or unable to participate
* Contraindication to adhesive placement, eg, epidermolysis bullosa
* Cancellation of the subject's planned CPET procedure.
* Tracheostomy tube presence (this will prevent proper placement of impedance cardiogram lead)

Ages: 7 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will enroll participants scheduled to undergo clinically indicated CPET procedures.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Autonomic data respiratory sinus arrhythmia among patients with chest pain | Data collected throughout cardiopulmonary exercise testing. Up to 90 minutes.
  Subjects will wear an ambulatory monitor during testing
Autonomic data respiratory sinus arrhythmia among patients with syncope | Data collected throughout cardiopulmonary exercise testing. Up to 90 minutes.
  Subjects will wear an ambulatory monitor during testing
Autonomic data respiratory sinus arrhythmia among patients post heart transplant | Data collected throughout cardiopulmonary exercise testing. Up to 90 minutes.
  Subjects will wear an ambulatory monitor during testing

CONTACTS AND LOCATIONS:
Overall Officials: Pornswan Ngamprasertwong, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Akselrod S, Gordon D, Ubel FA, Shannon DC, Berger AC, Cohen RJ. Power spectrum analysis of heart rate fluctuation: a quantitative probe of beat-to-beat cardiovascular control. Science. 1981 Jul 10;213(4504):220-2. doi: 10.1126/science.6166045.
- [Background] Dahlqvist JA, Karlsson M, Wiklund U, Hornsten R, Stromvall-Larsson E, Berggren H, Hanseus K, Johansson S, Rydberg A. Heart rate variability in children with Fontan circulation: lateral tunnel and extracardiac conduit. Pediatr Cardiol. 2012 Feb;33(2):307-15. doi: 10.1007/s00246-011-0126-2. Epub 2011 Oct 8. PMID 21984213
- [Background] Grossman P, van Beek J, Wientjes C. A comparison of three quantification methods for estimation of respiratory sinus arrhythmia. Psychophysiology. 1990 Nov;27(6):702-14. doi: 10.1111/j.1469-8986.1990.tb03198.x. PMID 2100356
- [Background] Grossman P, Taylor EW. Toward understanding respiratory sinus arrhythmia: relations to cardiac vagal tone, evolution and biobehavioral functions. Biol Psychol. 2007 Feb;74(2):263-85. doi: 10.1016/j.biopsycho.2005.11.014. Epub 2006 Nov 1. PMID 17081672
- [Background] Vinik AI, Ziegler D. Diabetic cardiovascular autonomic neuropathy. Circulation. 2007 Jan 23;115(3):387-97. doi: 10.1161/CIRCULATIONAHA.106.634949. No abstract available. PMID 17242296
- [Background] Harteveld LM, Nederend I, Ten Harkel ADJ, Schutte NM, de Rooij SR, Vrijkotte TGM, Oldenhof H, Popma A, Jansen LMC, Suurland J, Swaab H, de Geus EJC; FemNAT-CD collaborators *. Maturation of the Cardiac Autonomic Nervous System Activity in Children and Adolescents. J Am Heart Assoc. 2021 Feb 16;10(4):e017405. doi: 10.1161/JAHA.120.017405. Epub 2021 Feb 2. PMID 33525889
- [Background] Willemsen GH, De Geus EJ, Klaver CH, Van Doornen LJ, Carroll D. Ambulatory monitoring of the impedance cardiogram. Psychophysiology. 1996 Mar;33(2):184-93. doi: 10.1111/j.1469-8986.1996.tb02122.x. PMID 8851246
- [Background] Saklani P, Krahn A, Klein G. Syncope. Circulation. 2013 Mar 26;127(12):1330-9. doi: 10.1161/CIRCULATIONAHA.112.138396. No abstract available. PMID 23529534
- [Background] Sheldon RS, Grubb BP 2nd, Olshansky B, Shen WK, Calkins H, Brignole M, Raj SR, Krahn AD, Morillo CA, Stewart JM, Sutton R, Sandroni P, Friday KJ, Hachul DT, Cohen MI, Lau DH, Mayuga KA, Moak JP, Sandhu RK, Kanjwal K. 2015 heart rhythm society expert consensus statement on the diagnosis and treatment of postural tachycardia syndrome, inappropriate sinus tachycardia, and vasovagal syncope. Heart Rhythm. 2015 Jun;12(6):e41-63. doi: 10.1016/j.hrthm.2015.03.029. Epub 2015 May 14. No abstract available. PMID 25980576
- [Background] Bottasso E. Toward the Existence of a Sympathetic Neuroplasticity Adaptive Mechanism Influencing the Immune Response. A Hypothetical View-Part I. Front Endocrinol (Lausanne). 2019 Sep 20;10:632. doi: 10.3389/fendo.2019.00632. eCollection 2019. PMID 31616373
- [Background] Bottasso E. Toward the Existence of a Sympathetic Neuroplasticity Adaptive Mechanism Influencing the Immune Response. A Hypothetical View-Part II. Front Endocrinol (Lausanne). 2019 Sep 18;10:633. doi: 10.3389/fendo.2019.00633. eCollection 2019. PMID 31620088